CLINICAL TRIAL: NCT04993404
Title: Study To Evaluate The Pharmacokinetics Of Jaktinib Hydrochloride Tablets In Subjects With Hepatic Impairment And Normal Hepatic Function
Brief Title: Pharmacokinetics Of Jaktinib In Subjects With Hepatic Impairment And Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK021
Record Dates: First submitted 2021-07-23; First posted 2021-08-06 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Hepatic Insufficiency; Healthy Subjects
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A：Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment (Child-Pugh Class A, score of 5 to 6, inclusive) will be administered a single dose of Jaktinib Hydrochloride Tablets.
  Interventions: Drug: Jaktinib Hydrochloride Tablets
- Cohort B：Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment (Child-Pugh Class B, score of 7 to 9, inclusive) will be administered a single dose of Jaktinib Hydrochloride Tablets.
  Interventions: Drug: Jaktinib Hydrochloride Tablets
- Cohort C：Normal Hepatic Function (Experimental): Participants with normal hepatic function matched to participants with hepatic impairment in Cohorts A and B (matched with regards to age, sex, body mass index) will be administered a single oral dose of Jaktinib Hydrochloride Tablets.
  Interventions: Drug: Jaktinib Hydrochloride Tablets
- Cohort D：Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment (Child-Pugh Class C, score of 10 to 11, inclusive) will be administered a single dose of Jaktinib Hydrochloride Tablets.
  Interventions: Drug: Jaktinib Hydrochloride Tablets

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Tablets — A single oral dose of 100 mg Jaktinib Hydrochloride Tablets will be administered.
  Other Names: Jaktinib

SUMMARY:
This multi-center, open-label, parallel-controlled, single-dose Phase 1 study is being conducted to directly characterize the pharmacokinetic (PK) profiles and safety of Jaktinib following administration of a single oral dose in subjects with varying degrees of hepatic impairment compared to healthy matched control subjects with normal hepatic function(matched by age, weight, and sex).

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an informed consent form. Ability to comply with trial and follow-up procedures.
* Age 18-79 years at the time of signing the ICF, either male or female.
* Male subjects body weight at least 50 kg, and female subjects body weight at least 45 kg. Body mass index (BMI) between 18 and 32 kg/m2 to participate.
* After physical examination, vital signs, laboratory examinations, 12-lead electrocardiogram examination, the investigator determined that it is suitable to participate in this study.
* Subjects are willing to take effective contraceptive measures from screening to 3 months after administration.

Additional Inclusion Criteria for Hepatic Impaired Subjects Only:

* Child-Pugh Clinical Assessment Score consistent with degree of hepatic impairment(Requires no use of albumin within 14 days), And it is dysfunction caused by previous primary liver disease.
* Any examination such as B-ultrasound, CT, MRI, FibroScan or liver biopsy confirms the presence of cirrhosis.

Additional Inclusion Criteria for Healthy Subjects Only:

* Have not taken any medicine within 2 weeks before administration; or have stable medication for at least 4 weeks before administration for the treatment of other comorbid diseases.

Exclusion Criteria:

* Drug-induced liver injury.
* Acute liver damage caused by various reasons.
* Patients with liver failure, or combined with dominant hepatic encephalopathy, liver cancer, etc., which the investigator believes are not suitable for participating in the study.
* Patients with a history of massive bleeding from esophageal varices without band ligation, sclerosing agent and TIPS treatment
* Subjects with suspected allergies to Jaktinib or its excipient.
* History of blood donation of 400 mL or more of blood within 3 months prior to screening.
* Drug dependency, a positive urine drug screen.
* Subjects with any significant clinical and laboratory abnormalities which may affect the safety evaluation.
* Subjects suffering from arrhythmia and requiring treatment, or QTcB > 480ms at screening.
* Subjects with clinical symptoms of active bacterial, viral, parasitic or fungal infections requiring treatment at screening.
* Subjects with known human immunodeficiency virus (HIV),
* Subjects with epilepsy or patients who have received psychotropic drug or sedatives during screening.
* Subjects who had experienced malignant tumors within the past 5 years (except for adequately treated local basal cell carcinoma of the skin and cervical carcinoma in situ that have been cured).
* Subjects who have participated in another clinical trial of a new drug or medical instrument within 3 months before screening.
* Females who are breastfeeding or pregnant at Screening.

Exclusion Criteria for Healthy Subjects Only:

* Subjects with hepatitis B surface antigen positive or HCV-RNA positive.
* Patients with a history of liver dysfunction, or physical examination and laboratory examination at screening indicate that there is or may have liver dysfunction.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]of Jaktinib and its metabolites（ZG0244 and ZG0245） | From day 1 to day 3
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Maximum Observed Plasma Concentration (Cmax) of Jaktinib and its metabolites（ZG0244 and ZG0245） | From day 1 to day 3
  To evaluate Maximum Observed Plasma Concentration (Cmax) of Jaktinib and its metabolites（ZG0244 and ZG0245）
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of Jaktinib and its metabolites（ZG0244 and ZG0245） | From day 1 to day 3
  The AUC (0-infinity) is the area under the plasma Jaktinib and its metabolites（ZG0244 and ZG0245）concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z)

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (7 days after dose administration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University; Weifeng Zhao, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

REFERENCES:
- [Derived] Zhao M, Zhang H, Ma S, Gong S, Wei C, Miao L, Zhao W. Clinical pharmacokinetic characteristics of Jaktinib in subjects with hepatic impairment in a phase I trial. Drug Metab Pharmacokinet. 2024 Dec;59:101030. doi: 10.1016/j.dmpk.2024.101030. Epub 2024 Jul 20. PMID 39442386